CLINICAL TRIAL: NCT07088874
Title: Novel Biomarkers to Predict Acute Kidney Injury and Chronic Kidney Disease After Radical Nephrectomy: an Exploratory Prospective Cohort Study
Brief Title: Novel Biomarkers and Postoperative Kidney Injury in Radical Nephrectomy
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, Qiongfang Wu, Peking University First Hospital, Peking University First Hospital
Other Study IDs: 2025-067
Record Dates: First submitted 2025-07-10; First posted 2025-07-28 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Nephrectomy; Acute Kidney Injury; Biomarker
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — perioperative AKI damaging (such as NGAL), stressful (such as TIMP-2, IGFBP-7) and functional novel (cystatin C) biomarkers and serum creatinine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AKI group/CKD group: 1. patients diagnosed with AKI after radical nephrectomy.
  2. patients diagnosed with the new onset/worsening of CKD after radical nephrectomy.
- non-AKI group/non-CKD group: 1. patients without AKI after radical nephrectomy.
  2. patients without new onset/worsening of CKD after radical nephrectomy.

SUMMARY:
The incidence of acute kidney injury (AKI) after radical nephrectomy exceeds 40%. Currently, the KDIGO criteria are the recognized diagnostic standard for AKI. These criteria primarily use serum creatinine and urine output as key indicators, but both parameters have certain limitations, such as delayed response, insensitivity, and inaccuracy. This study aims to simultaneously monitor perioperative novel renal damaging, stressful, and functional biomarkers in patients undergoing radical nephrectomy, and to investigate their predictive value for AKI and postoperative 1-year chronic kidney disease (CKD).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Scheduled to undergo unilateral radical nephrectomy.

Exclusion Criteria:

* Solitary kidney;
* Preoperative diagnosis of chronic kidney disease stages G4 or G5 (GFR <30 mL/min/1.73m²);
* Tumor invasion of the vena cava requiring thrombectomy;
* Other conditions deemed by the investigator as unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Targeting patients undergoing radical nephrectomy for renal cell carcinoma
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-02 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
The urinary [TIMP-2]×[IGFBP-7], urinary NGAL, urinary KIM-1, serum cystatin C and their combinations to predict postoperative AKI occurring within 7 days. | Up to 7 days after surgery.
  Novel biomarkers above were collected at the end of surgery, and at postoperative 1h, 6h, and 20h. AKI diagnosed according to 2012 KDIGO criteria (occurring within 7 days after surgery).

SECONDARY OUTCOMES:
The urinary [TIMP-2]×[IGFBP-7], urinary NGAL, urinary KIM-1, serum cystatin C and their combinations to predict new onset/worsening CKD occurring within 1 year after surgery. | Up to 1 year after surgery
  Novel biomarkers above were collected before and at the end of surgery, and at postoperative 1h, 6h, and 20h. CKD diagnosed according to 2024 KDIGO-CKD criteria (occurring within 1 year after surgery).
The urinary [TIMP-2]×[IGFBP-7], urinary NGAL, urinary KIM-1, serum cystatin C combined with clinically important risk factors to predict postoperative AKI occurring within 7 days after surgery. | Up to 7 days after surgery.
  Novel biomarkers above were collected before and at the end of surgery, and at postoperative 1h, 6h, and 20h. AKI diagnosed according to 2012 KDIGO criteria (occurring within 7 days after surgery).
The postoperative urinary [TIMP-2]×[IGFBP-7], urinary NGAL, urinary KIM-1, serum cystatin C combined with clinically important risk factors to predict postoperative the new onset/worsening CKD occurring within 1 year after surgery. | Up to 1 year after surgery.
  Novel biomarkers above were collected before and at the end of surgery, and at postoperative 1h, 6h, and 20h. CKD diagnosed according to 2024 KDIGO-CKD criteria (occurring within 1 year after surgery).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Critical Care Medicine, Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Antonelli A, Allinovi M, Cocci A, Russo GI, Schiavina R, Rocco B, Giovannalberto P, Celia A, Galfano A, Varca V, Bozzini G, Ceruti C, Greco F, Verze P, Pastore AL, Porreca A, Minervini A; AGILE Group. The Predictive Role of Biomarkers for the Detection of Acute Kidney Injury After Partial or Radical Nephrectomy: A Systematic Review of the Literature. Eur Urol Focus. 2020 Mar 15;6(2):344-353. doi: 10.1016/j.euf.2018.09.020. Epub 2018 Oct 9. PMID 30309817
- [Background] Rossiter A, La A, Koyner JL, Forni LG. New biomarkers in acute kidney injury. Crit Rev Clin Lab Sci. 2024 Jan;61(1):23-44. doi: 10.1080/10408363.2023.2242481. Epub 2023 Sep 5. PMID 37668397
- [Background] Ostermann M, Zarbock A, Goldstein S, Kashani K, Macedo E, Murugan R, Bell M, Forni L, Guzzi L, Joannidis M, Kane-Gill SL, Legrand M, Mehta R, Murray PT, Pickkers P, Plebani M, Prowle J, Ricci Z, Rimmele T, Rosner M, Shaw AD, Kellum JA, Ronco C. Recommendations on Acute Kidney Injury Biomarkers From the Acute Disease Quality Initiative Consensus Conference: A Consensus Statement. JAMA Netw Open. 2020 Oct 1;3(10):e2019209. doi: 10.1001/jamanetworkopen.2020.19209. PMID 33021646
- [Background] Gocze I, Jauch D, Gotz M, Kennedy P, Jung B, Zeman F, Gnewuch C, Graf BM, Gnann W, Banas B, Bein T, Schlitt HJ, Bergler T. Biomarker-guided Intervention to Prevent Acute Kidney Injury After Major Surgery: The Prospective Randomized BigpAK Study. Ann Surg. 2018 Jun;267(6):1013-1020. doi: 10.1097/SLA.0000000000002485. PMID 28857811
- [Background] Kane-Gill SL, Peerapornratana S, Wong A, Murugan R, Groetzinger LM, Kim C, Smithburger PL, Then J, Kellum JA. Use of tissue inhibitor of metalloproteinase 2 and insulin-like growth factor binding protein 7 [TIMP2]*[IGFBP7] as an AKI risk screening tool to manage patients in the real-world setting. J Crit Care. 2020 Jun;57:97-101. doi: 10.1016/j.jcrc.2020.02.002. Epub 2020 Feb 4. PMID 32086072
- [Background] Leem AY, Park MS, Park BH, Jung WJ, Chung KS, Kim SY, Kim EY, Jung JY, Kang YA, Kim YS, Kim SK, Chang J, Song JH. Value of Serum Cystatin C Measurement in the Diagnosis of Sepsis-Induced Kidney Injury and Prediction of Renal Function Recovery. Yonsei Med J. 2017 May;58(3):604-612. doi: 10.3349/ymj.2017.58.3.604. PMID 28332367
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) CKD Work Group. KDIGO 2024 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease. Kidney Int. 2024 Apr;105(4S):S117-S314. doi: 10.1016/j.kint.2023.10.018. No abstract available. PMID 38490803